CLINICAL TRIAL: NCT05333822
Title: Effects of Bashan,a Vegetable Plant Based Compound Drink , on Glucose in Type 2 Diabetes Patients and Its Related Mechanisms
Brief Title: Effects of Bashan on Glucose in Type 2 Diabetes Patients and Its Related Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Zilin Sun, Professor, Zhongda Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Bashan-01
Record Dates: First submitted 2022-03-31; First posted 2022-04-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; glucose; TIR
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bashan (Experimental): a vegetable plant based compound drink add after three meals for 14 days
  Interventions: Dietary Supplement: Bashan
- Water (Placebo Comparator): water as placebo
  Interventions: Other: water

INTERVENTIONS:
Dietary Supplement: Bashan — a vegetable plant based compound drink add after three meals for 14 days
  Arms: Bashan
Other: water — water as placebo
  Arms: Water

SUMMARY:
The study aimed to observe the effect of targeted diet on blood glucose improvement in type 2 diabetic patients by continuous glucose monitoring and to explore the possible mechanism of targeted diet on blood glucose improvement in type 2 diabetic patients.

DETAILED DESCRIPTION:
Subjects were studied on 2 occasions, separated by at least 7 days, in a randomized fashion. The order of the enteral infusions was randomized and facilitated by a biostatistician who generated the randomization code and a research officer who prepared the study solutions, but were not involved in data collection or analysis. Each occasion would last for 14 days maintaining daily eating habits without intervention and take 180ml mineral water or Bashan three times a day after meals. During the 2-week test, all subjects will still wear continuous glucose monitoring systems. Before and after the intervention, the standard meal test would be carried out on the subjects, and the samples of serum and feces, etc. of the subjects would be collected for the following tests.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes;
2. With only diet and exercise control for at least 3 months or stable use of basal insulin for hypoglycemic treatment for at least 3 months;
3. Fasting blood glucose is greater than 7.0mmol/L, 2h postprandial blood glucose is greater than 11.1mmol/L, and glycosylated glycoprotein is 7.0-8.5%;
4. 18-60 years old;
5. Those who have voluntarily signed the informed consent.

Exclusion Criteria:

1. Pregnant or lactating women or women planning pregnancy who are unwilling to take or do not take adequate contraceptive measures;
2. Drinking (more than 5 times a week, and 100g liquor or 250g yellow wine or 5 bottles of beer above on average each time) or smoking history;
3. Serious mental illness in the past 6 months;
4. Those who have undergone gastrointestinal surgery, except appendicitis and hernia surgery;
5. Patients with chronic or persistent hepatitis, patients with severe liver disease such as cirrhosis, or those whose hepatitis B surface antigen (HBsAg) is positive and is accompanied by abnormal liver function (serum glutamic pyruvic transaminase and aspartate aminotransferase are 2.5 times the normal value).
6. Suffering from Cushing's syndrome, pituitary dysfunction and other endocrine system diseases;
7. Factors that hinder participation in the research, such as unstable medical conditions, including blood pressure and cardiovascular disease, etc.

   i. malignant hypertension (blood pressure > 180/110mmHg, systolic blood pressure > 180mmHg or diastolic blood pressure > 110mmHg); unstable blood pressure control; ii. myocardial infarction, other acute cardiac events requiring hospitalization, stroke, transient ischemic attack, or treatment of acute congestive heart failure;
8. Suffering from infectious diseases such as tuberculosis and AIDS;
9. Anemia: hemoglobin < 10g/dl;
10. Severe renal insufficiency: GFR ≤ 30ml/min/1.73m2;
11. Ketosis, ketoacidosis and uncontrolled infection in recent 1 month;
12. Those who are deemed unsuitable for participating in this clinical trial by the researcher for any reason;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
blood glucose improvement in type 2 diabetic patients by continuous glucose monitoring. | 14 days

SECONDARY OUTCOMES:
insulin C-peptide gastric emptying | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Zilin Sun, Study Chair — Zhongda Hospital
Locations (1):
- Department of Endocrinology, Zhongda Hospital. Institute of Diabetes, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The study didn't plan to share the data

REFERENCES:
- [Background] Zhou M, Astell-Burt T, Bi Y, Feng X, Jiang Y, Li Y, Page A, Wang L, Xu Y, Wang L, Zhao W, Ning G. Geographical variation in diabetes prevalence and detection in china: multilevel spatial analysis of 98,058 adults. Diabetes Care. 2015 Jan;38(1):72-81. doi: 10.2337/dc14-1100. Epub 2014 Oct 28. PMID 25352654
- [Background] Ji X, Leng XY, Dong Y, Ma YH, Xu W, Cao XP, Hou XH, Dong Q, Tan L, Yu JT. Modifiable risk factors for carotid atherosclerosis: a meta-analysis and systematic review. Ann Transl Med. 2019 Nov;7(22):632. doi: 10.21037/atm.2019.10.115. PMID 31930033
- [Background] Karagodin VP, Sukhorukov VN, Orekhov AN, Yet SF, Sobenin IA. Atherosclerosis prevention: the role of special diets and functional food. Front Biosci (Elite Ed). 2020 Jan 1;12(1):95-101. doi: 10.2741/E859. PMID 31585871
- [Background] Post RE, Mainous AG 3rd, King DE, Simpson KN. Dietary fiber for the treatment of type 2 diabetes mellitus: a meta-analysis. J Am Board Fam Med. 2012 Jan-Feb;25(1):16-23. doi: 10.3122/jabfm.2012.01.110148. PMID 22218620
- [Background] Legeay S, Rodier M, Fillon L, Faure S, Clere N. Epigallocatechin Gallate: A Review of Its Beneficial Properties to Prevent Metabolic Syndrome. Nutrients. 2015 Jul 7;7(7):5443-68. doi: 10.3390/nu7075230. PMID 26198245
- [Background] Li K, Yao F, Xue Q, Fan H, Yang L, Li X, Sun L, Liu Y. Inhibitory effects against alpha-glucosidase and alpha-amylase of the flavonoids-rich extract from Scutellaria baicalensis shoots and interpretation of structure-activity relationship of its eight flavonoids by a refined assign-score method. Chem Cent J. 2018 Jul 12;12(1):82. doi: 10.1186/s13065-018-0445-y. PMID 30003449
- [Background] Gu Y, Wang X, Li J, Zhang Y, Zhong H, Liu R, Zhang D, Feng Q, Xie X, Hong J, Ren H, Liu W, Ma J, Su Q, Zhang H, Yang J, Wang X, Zhao X, Gu W, Bi Y, Peng Y, Xu X, Xia H, Li F, Xu X, Yang H, Xu G, Madsen L, Kristiansen K, Ning G, Wang W. Analyses of gut microbiota and plasma bile acids enable stratification of patients for antidiabetic treatment. Nat Commun. 2017 Nov 27;8(1):1785. doi: 10.1038/s41467-017-01682-2. PMID 29176714
- [Background] Chen C, Zeng Y, Xu J, Zheng H, Liu J, Fan R, Zhu W, Yuan L, Qin Y, Chen S, Zhou Y, Wu Y, Wan J, Mi M, Wang J. Therapeutic effects of soluble dietary fiber consumption on type 2 diabetes mellitus. Exp Ther Med. 2016 Aug;12(2):1232-1242. doi: 10.3892/etm.2016.3377. Epub 2016 May 20. PMID 27446349
- [Background] Fan J, Johnson MH, Lila MA, Yousef G, de Mejia EG. Berry and Citrus Phenolic Compounds Inhibit Dipeptidyl Peptidase IV: Implications in Diabetes Management. Evid Based Complement Alternat Med. 2013;2013:479505. doi: 10.1155/2013/479505. Epub 2013 Aug 29. PMID 24069048